CLINICAL TRIAL: NCT02112357
Title: FOrMAT - Feasibility of a Molecular Characterisation Approach to Treatment
Brief Title: Feasibility of a Molecular Characterisation Approach to Treatment
Acronym: FOrMAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 3994
Record Dates: First submitted 2014-03-31; First posted 2014-04-11 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Advanced Gastrointestinal Cancers
Keywords: molecular profiling; genetic sequencing; personalised medicine; gastrointestinal cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Both fresh frozen tissue and formalin-fixed paraffin-embedded (FFPE) tumour samples will be obtained.
  Biopsies may be taken at entry to the study and/or at the time of radiological response assessment. Each patient can have a maximum of 3 research biopsies in this study.
  Up to 35 ml of blood will be collected at study entry to provide normal germline DNA and for possible additional biomarker analysis. If the patient has consented to optional blood sample collection, then additional blood samples will also be collected at the time of radiological response assessment to study molecular changes that occur during treatment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Targeted genetic sequencing of tumour specimen

SUMMARY:
This study will assess the feasibility of sequencing locally advanced/metastatic gastrointestinal cancers in real-time to enable future treatment stratification by molecular characteristics. Targeted next generation sequencing of a panel of genes will be performed on tumour specimens and results will be discussed at a Sequencing Tumour Board to establish if a patient is potentially suitable for a targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic gastrointestinal cancer (including oesophageal, oesophagogastric junction, gastric, pancreatic, biliary and colorectal cancers).
2. Histological or cytological confirmation of diagnosis of malignancy.
3. Patients must either:

   1. Have received at least one line of treatment for locally advanced/metastatic disease OR
   2. Be about to start/currently undergoing their first line of treatment for locally advanced/metastatic disease
4. 18 years of age and over .
5. Performance status less than or equal to 2.
6. Able to provide fully informed consent.
7. Patients must either:

   1. Have an available tumour specimen (FFPE or fresh frozen) from either the primary tumour or a metastasis. Metastatic samples may be from any site with the exception of bone. OR
   2. Have a site of disease which is amendable to biopsy

Exclusion Criteria:

* There are no specific exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced or metastatic gastrointestinal cancer (including gastroesophageal, pancreatic, biliary tract and colorectal cancer)
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients in whom a currently actionable molecular alteration was detected by genetic sequencing. | 18 months

SECONDARY OUTCOMES:
The concordance of results obtained from genetic sequencing compared to standard clinically validated techniques. | 18 months
The proportion of patients in whom genetic sequencing was successfully performed. | 18 months
The percentage of patients with a currently actionable genetic alteration who received targeted therapy as a result of genetic sequencing. | 18 months
  To assess the potential impact of genetic sequencing results on patients' treatment
Evaluation of the time required to obtain genetic sequencing results to see if genetic sequencing could be practically incorporated into clinical practice. | 18 months
  To assess whether genetic sequencing results can be obtained within a clinically meaningful timeframe
The proportion of screened patients who decide to participate in the trial and their reasons for participation or deciding not to participate. | 18 months
The concordance of results obtained from core biopsy versus fine needle aspirate specimens from individual patients. | 18 months
The number needed to enroll into the trial to identify one patient with a targetable genetic alteration and the number needed to enroll into the trial to treat one patient with a targeted agent. | 18 months

OTHER OUTCOMES:
Response rate for patients who received a targeted treatment as a result of genetic sequencing. | 18 months
Overall survival of patients who received targeted treatment. | 18 months
Evaluation of any changes in molecular markers at the time of disease progression or response to those from previous specimens. | 18 months
  To examine tumour heterogeneity in patients with paired specimens
Description of the microRNA expression profile of gastrointestinal tumours | 18 months
Evaluation of any changes in circulating tumour DNA at the time of progression or response in comparison to previous specimens | 18 months
Duration of response for patients who received a targeted treatment as a result of genetic sequencing. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Naureen Starling, BSc, MBBS, MRCP, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London and Surrey, United Kingdom

REFERENCES:
- [Derived] Mansukhani S, Barber LJ, Kleftogiannis D, Moorcraft SY, Davidson M, Woolston A, Proszek PZ, Griffiths B, Fenwick K, Herman B, Matthews N, O'Leary B, Hulkki S, Gonzalez De Castro D, Patel A, Wotherspoon A, Okachi A, Rana I, Begum R, Davies MN, Powles T, von Loga K, Hubank M, Turner N, Watkins D, Chau I, Cunningham D, Lise S, Starling N, Gerlinger M. Ultra-Sensitive Mutation Detection and Genome-Wide DNA Copy Number Reconstruction by Error-Corrected Circulating Tumor DNA Sequencing. Clin Chem. 2018 Nov;64(11):1626-1635. doi: 10.1373/clinchem.2018.289629. Epub 2018 Aug 27. PMID 30150316
- [Derived] Moorcraft SY, Gonzalez de Castro D, Cunningham D, Jones T, Walker BA, Peckitt C, Yuan LC, Frampton M, Begum R, Eltahir Z, Wotherspoon A, Teixeira Mendes LS, Hulkki Wilson S, Gillbanks A, Baratelli C, Fotiadis N, Patel A, Braconi C, Valeri N, Gerlinger M, Rao S, Watkins D, Chau I, Starling N. Investigating the feasibility of tumour molecular profiling in gastrointestinal malignancies in routine clinical practice. Ann Oncol. 2018 Jan 1;29(1):230-236. doi: 10.1093/annonc/mdx631. PMID 29361134